CLINICAL TRIAL: NCT03256565
Title: Correlation Between Q-tip Test and Urodynamic Study in Women With Stress Urinary Incontinence
Brief Title: Q-tip Test and Urodynamic Study
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 106060-E
Record Dates: First submitted 2017-08-13; First posted 2017-08-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Q-tip test — A Q-Tip lubricated with anesthetic gel is inserted into the urethra, woman is then asked to cough and strain, and the angle of the Q-tip rotates is recorded.

SUMMARY:
Urethral hypermobility, which can be assessed with Q-tip test, has been considered to be partly responsible for pathogenesis of women with stress urinary incontinence (SUI). Nonetheless, Q-tip test has lost favor due to patient discomfort. Thus, the purpose of this study was to search a surrogate for assessment of urethral hypermobility by correlating the Q-tip angle and the urodynamic variables in women with SUI.

DETAILED DESCRIPTION:
All women with SUI and underwent Q-tip testing were reviewed. Patient characteristics, degree of prolapse determined by Pelvic Organ Prolapse Quantification system, Q-tip angle, the results of urodynamic studies, the Urinary Distress Inventory (UDI-6) Questionnaire and Incontinence Impact (IIQ-7) Questionnaire were reviewed from their medical records. Spearman correlation test, and univariate and multivariate backward stepwise linear regression analysis were performed as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* all women with stress urinary incontinence, who underwent both Q-tip testing and urodynamic study, and completed the Urinary Distress Inventory (UDI-6) Questionnaire and Incontinence Impact (IIQ-7) Questionnaire

Exclusion Criteria:

* women who had incomplete exam or questionnaires

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Correlations of Q-tip angle with pressure transmission ratio | Between 2014 and 2020
  Correlations of Q-tip angle with pressure transmission ratio at maximum urethral pressure during stress urethral pressure profile testing

SECONDARY OUTCOMES:
Correlations of Q-tip angle with the other parameters of urodynamic studies | Between 2014 and 2020
  clinical and urodynamic variables include maximum flow rate, voided volume, post-void residual, voiding time, strong desire, PdetQmax, MUCP, functional profile length
Correlations of Q-tip angle with pad weight | Between 2014 and 2020
  Correlations of Q-tip angle with 20 min pad testing result
Correlations of Q-tip angle with symptoms | Between 2014 and 2020
  Correlations of Q-tip angle with questionnaires of urinary symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided